CLINICAL TRIAL: NCT05081271
Title: COVID-19 Booster Vaccination in Persons With Multiple Sclerosis
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Most potential participants had already received their booster vaccinations outside of the study
Sponsor: Griffin Hospital (Other)
Collaborators: Yale-Griffin Prevention Research Center (Other); Multiple Sclerosis Treatment Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12
Record Dates: First submitted 2021-10-14; First posted 2021-10-18 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The proposed pilot study is a prospective, randomized open label study with two treatment assignments: one group will receive a homologous booster vaccine and the other a heterologous booster vaccine.
Masking Description: Open label study. No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Homologous booster vaccine group (Active Comparator): A single dose booster of the same type of COVID-19 vaccine (i.e., mRNA or DNA) that the study participant received as part of an initial vaccine series prior to enrolling in this study.
  Interventions: Biological: Homologous booster
- Heterologous booster vaccine group (Active Comparator): A single dose booster of the opposite type of COVID-19 vaccine (i.e., mRNA or DNA) that the study participant received as part of an initial vaccine series prior to enrolling in this study.
  Interventions: Biological: Heterologous booster

INTERVENTIONS:
Biological: Homologous booster — Group 1 will receive a booster dose of a homologous vaccine and Group 2 a heterologous vaccine. This means Ad26.COV2.S if they originally received BNT162b2 or mRNA-1273 or vice versa
  Arms: Homologous booster vaccine group
Biological: Heterologous booster — Group 1 will receive a booster dose of a homologous vaccine and Group 2 a heterologous vaccine. This means Ad26.COV2.S if they originally received BNT162b2 or mRNA-1273 or vice versa
  Arms: Heterologous booster vaccine group

SUMMARY:
The success of the U.S. vaccination program against SARS-Cov-2 is shown by a dramatic drop in infection rates, hospitalizations and deaths.However, it appears that many persons who take medications that chronically suppress the immune system do not produce neutralizing antibodies to COVID-19 proteins in response to vaccination. This group includes a significant number of persons with multiple sclerosis (PWMS), many of whom are on therapies that chronically suppress their immune function. It is unclear what advice clinicians should provide regarding COVID-19 precautions to patients who fail to develop detectable COVID-19 spike protein antibodies using standard commercially-available tests after a standard series of vaccination, or whether they should test for antibody responses to COVID-19 vaccines in the absence of guidelines. A key research question is whether, in the absence of stopping or reducing potentially immune-altering therapies, there is a way to increase the likelihood of a neutralizing antibody response to COVID-19 vaccination in PWMS who are taking immune suppressive medications.

DETAILED DESCRIPTION:
The goal of this study is to test whether adding booster doses of COVID-19 vaccine to PWMS can improve the immune response to COVID-19.

Specific Aims:

* To compare pre and post anti-COVID-19 immunity after a booster vaccination in PWMS who initially test negative for neutralizing antibodies to COVID-19 after initial vaccination;
* To determine how disease modifying treatments, baseline antibody panels and lymphocyte subsets associate with the efficacy of booster vaccines;
* To compare immune responses between homologous vs. heterologous booster vaccination.

Research Implications:

It is hoped that the results of this study will help guide clinical recommendations on the use of booster vaccination and whether to endorse heterologous versus homologous boosters. It is also hoped that this study will add to the growing body of data on COVID-19 immunity after vaccination in PWMS on various disease modifying treatments (DMTs).

Hypotheses:

* Booster doses of COVID-19 vaccines will improve antibody-based immunity to COVID-19in PWMS who initially test negative for neutralizing antibodies to COVID-19 after initial vaccination;
* This boost in immunity will occur irrespective of disease modifying therapy (DMT);
* Heterologous prime-boost combinations will show greater immune responses than homologous prime-boost combinations.

Background:

Multiple Sclerosis (MS) is an autoimmune condition associated with focal inflammatory infiltrates in the brain consisting of T and B lymphocytes, macrophages and activated microglial cells, with the principal target being the myelin sheath of central nervous system (CNS) axons. The approach to treating MS involves disease-modifying therapies (DMT) that have the effect of reducing access of potentially myelin-autoreactive immune cells to the CNS compartment. These treatments are shown to reduce exacerbations of disease and, to some degree, delay progression of neurological disability, both by clinical assessment, and, by the best surrogate marker to date, magnetic resonance imaging of the brain.

DMTs used to treat MS target adaptive immune responses in various ways. These include medications that shift cytokine and lymphocyte subsets towards less inflammatory activity, interfere with trafficking of lymphocytes in the circulation or central nervous system, or otherwise inhibit lymphocytes through nonspecific or subset depletion.

Approved and off-label treatments for MS include:

1. anti-CD20 (CD20 is a B lymphocyte receptor) monoclonal antibodies (ocrelizumab, rituximab and ofatunumab);
2. lymphocyte-sequestering drugs (fingolimod, onzanimod, siponomod);
3. adhesion molecule antibodies that prevent CNS lymphocyte trafficking(natalizumab);
4. nuclear erythroid 2-related factor two (Nrf2) modulators (dimethyl fumarate, diroxmel fumarate);
5. nonselective lymphocyte-depleters (cyclophosphamide, cladribine, alemtuzumab);
6. replication blocking lymphostatic drugs (teriflunomide) and immune modulators (interferon, glatiramer acetate).

All of these mechanisms could, theoretically, influence immune responses to vaccination. Live or live attenuated vaccines are contraindicated with several DMTs due to the risk of immune suppression. For COVID-19 immunity, both B and T lymphocyte activation is important. DMTs that are more immune-suppressive have shown attenuated responses to influenza vaccines and, presumably, would show the same for COVID-19 vaccines. These include the lymphocyte-sequestering drugs (e.g., fingolimod, onzanimod and siponimod), the antiCd20+ depleting drugs (e.g., ocrelizumab, ofatunumab and rituximab), and the general immune suppressants (e.g., alemtuzumab or cladribine). DMTs that have not been shown to inhibit immune responses to influenza vaccines include the interferons, glatiramer acetate, dimethyl fumarates, diroximel, and teriflunomide.

Currently three COVID-19 vaccines in the U.S. have either been approved for use or granted Emergency Use Authorization by the U.S. Food and Drug Administration (FDA). BNT162b2, manufactured by Pfizer, Inc. and BioNTech, Inc. and mRNA-1273, manufactured by Moderna, Inc., are RNA-based vaccines. They consist of modified COVID-19 mRNA sequences for the receptor-binding domain (RBD) of the M-spike protein. The mRNAs enter host cells via a lipid nanoparticle delivery system, where they are transcribed by host cell enzymes to produce a stabilized prefusion SARS-CoV-2 spike protein (S-2P), which localizes to the cell surface and presented as antigen for the host immune system. Ad26.COV2.S, manufactured by Johnson & Johnson/Janssen, is a dsDNA vaccine that employs a similar strategy, the difference being that it enters the host cell nucleus via a non-replicating adenovirus vector, where it is transcribed to make spike protein.

In some literature reviews and studies, PWMS, including those on a wide spectrum of DMTs, do not seem to be at greater risk per se of increased morbidity and mortality from COVID-19 infection. A review of 873 published cases of COVID-19 multiple sclerosis patients, found that the overall mortality rate was 4% and that an additional 3% required some form of ventilation. Furthermore, immune suppressive treatments did not appear to be a risk factor for severe disease. An unfavorable prognosis for 28 PWMS who contracted COVID-19 in a Spanish study was related to older age and greater disability. These and other observations have prompted some to speculate that relative immune suppression may actually protect PWMS against inflammatory storm that accompanies severe COVID-19 infection. On the other hand, a meta-analysis of 84 reports of PWMS with COVID-19 infection and their DMT treatments, while not finding a relationship between the type of DMT and COVID-19 course, did find that the highest mortality rate, e.g., 4% out of a 1.8% overall mortality rate of those infected, was in persons treated with rituximab, a monoclonal antibody that suppresses B lymphocytes and antibody production. This higher incidence of severe COVID-19 infection in MS patients on rituximab was confirmed by another retrospective study. A similar monoclonal antibody, ocrelizumab, was found to be associated with suppressed COVID-19 specific antibodies compared to other DMTs among 59 PWMS who had laboratory-confirmed COVID-19 infection. However, COVID-19 specific T lymphocyte assays were not different between ocrelizumab and other DMTs.

While there is a paucity of data relating to MS, DMTs and acquired immunity to COVID-19 infection, there is evidence that the use of some DMTs in MS can attenuate the immune response to various viral and nonviral vaccines. A number of DMTs in common use in MS patients increase their risk for a number of infectious complications, including bacterial and nonbacterial upper and lower respiratory tract infections, herpes virus infections, cryptococcal meningitis, progressive multifocal leukoencephalopathy and reactivation of latent tuberculosis and hepatitis B infections. Therefore, clinicians must be mindful of the initiation and timing of vaccinations, as well as the selection of DMTs in particular patients, to mitigate the risk of opportunistic infections.

This is critical with respect to assessing the protective effect of COVID-19 vaccination during the pandemic, especially as public health measures against COVID-19, e.g., social distancing, mask wearing, work and school restrictions, have been relaxed for vaccinated persons. What is clear from some preliminary studies is that PWMS on particular DMTs have attenuated responses to COVID-19 vaccines. Furthermore, there are approximately a dozen ongoing studies assessing the impact of DMTs on COVID-19 vaccination. One such study looked at antibody levels to the COVID-19 spike protein after vaccination with BNT162b2 in patients on no treatment or high efficacy DMTs, e.g., fingolimod, cladribine, or ocrelizumab. Humoral immunity in patients on ocrelizumab was achieved in 22.7%; fingolimod 3.8%, and cladribine 100% 33.

The potential attenuation of immunity to COVID-19 vaccination in PWMS at present is an unresolved dilemma for patients and physicians. Of course, this applies to other patients as well, including those on immune suppressive treatments for cancer or rheumatological diseases. There are commercially available assays to measure COVID-19 spike protein antibodies, but what are physicians to tell patients who test negative for these antibodies after vaccination. Some MS colleagues take the position that the tests should not be ordered due to a lack of guidance as to how to use that information.

One possible way to mitigate this dilemma is to administer booster vaccinations. A number of clinical investigators in other medical specialties are testing this approach. Indeed, since the extent to which the current vaccines induce long-term immunity to COVID-19 ia unknoqn, this is a relevant issue for the general population as well. A small study of 33 adults showed that high levels of antibodies persisted for six months after vaccination with mRNA-1273.

A booster vaccine may be homologous (same vaccine) or heterologous (different vaccine) relative to the initial vaccine. Evidence from one mouse study indicates that the immune response is more robust from heterologous combinations of mRNA and DNA COVID-19 vaccines than homologous combinations, particularly in the induction of T cells, which is believed to be more important for long term immunity. Another rationale for the use of heterologous combinations is to administer one dose each of the combination, rather than a full series of the mRNA vaccine, to determine which strategy produces more robust immunity.

This study will attempt to address whether giving a heterologous dose of a booster vaccine will increase the chance of both antibody production and T lymphocyte activation in PWMS who do not initially show evidence of antibody reactivity.

Research Plan:

The research team will recruit PWMS who have completed vaccination against COVID-19 and test negative for COVID-19 spike protein antibodies using a commercial assay. Subjects will have baseline blood drawn for T and B lymphocyte subsets, quantitative immune globulins and COVID-19 spike protein antibodies. Women of child-bearing potential will have a urine pregnancy test. Baseline, demographic and disease specific variables will be collected.

Subjects will be randomized on a stratified basis to one of two treatment groups: Group 1 will receive a booster dose of a homologous vaccine and Group 2 a heterologous vaccine. Depending on the initial vaccine series received, this means Ad26.COV2.S if they originally received BNT162b2 or mRNA-1273 or vice versa.

Subjects will return to the clinic 4 to 6 weeks later to be retested for COVID-19 spike protein antibodies. Reactions to the booster vaccine and any potential adverse events will be recorded.

Visit 1:

* Clinical screening; review of clinical course; medications; body mass index; vital signs; physical exam, neurological exam; and urine pregnancy test (if applicable);
* Phlebotomy for B and T lymphocyte subsets, quantitative immune globulins and COVID-19 spike antibodies;
* Administration of vaccine, followed by monitoring for any adverse effects for 15 to 30 minutes.

Visit 2:

* Physical and neurological examination
* Change of medications, assessment of disease activity (including relapses), adverse events including an assessment of relationship to vaccination
* Phlebotomy for COVID-19 spike protein antibodies

Data Analysis:

* Spike protein antibody titers, quantitative immune globulins, B & T cell subsets and COVID-specific T lymphocytes will be analyzed between Groups 1 & 2 and within Groups 1 & 2.
* DMT treatment, prior COVID-19 and/or vaccination history will be treated as covariates.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of clinically definite multiple sclerosis (CDMS) by the 2017 McDonald Criteria 38;
2. Age greater than or equal to 18 years;
3. Ability to travel to Griffin Hospital for phlebotomy and booster vaccination;
4. Completion of an initial COVID-19 vaccine series at least 4 weeks prior to booster randomization (i.e., two doses of either BNT162b2 or mRNA-1273, or one dose of Ad26.COV2.S);
5. Prior negative test for COVID-19 spike protein antibodies using a commercial assay;
6. Willing to undergo a booster vaccination with either BNT162b2, mRNA-1273 or Ad26.COV2.S.

Exclusion Criteria:

1. Inability to give consent;
2. Non-fluency in English;
3. Inability to adhere to the protocol;
4. Anticipated life expectancy of less than six months;
5. Lack of a primary care physician or treating neurologist;
6. Taking an immunosuppressive medication or chemotherapy for any other conditions aside fromMS;
7. Presence of another autoimmune condition requiring treatment;
8. Active treatment for cancer;
9. History of heavy alcohol use within the past year, as defined by the following criteria:

   1. Men: 5 or more alcoholic beverages per session or per day, or 15 or more per week;
   2. Women: 4 or more alcoholic beverages per session or per day, or 8 or more per week;
10. History of illicit drug abuse, e.g., cocaine, heroin, PCP, and/or narcotics within the past year;
11. Any condition that would jeopardize the safety or rights of the subject, make it unlikely for the subject to complete the study, or confound the study results.
12. Anaphylactic or other severe reaction to a previously administered COVID-19 vaccine;
13. MS relapse or worsening symptoms after initial COVID-19 vaccination.
14. Positive urine pregnancy test at screening [women only]. Test is waived in women who are post-menopausal or incapable of conception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Percent who test positive for COVID-19 spike protein antibodies following booster | 4-6 weeks
  Percentage of subjects who test positive for COVID-19 spike protein antibodies following a booster vaccination.

SECONDARY OUTCOMES:
Comparison of COVID-19 spike protein antibodies based on booster received | 4-6 weeks
  Comparison of percentage of subjects who test positive for COVID-19 specific spike protein antibodies between those who receive homologous vs. heterologous boosters from baseline;
Comparison of COVID-19 spike protein antibodies based on disease-modifying treatment | 4-6 weeks
  Comparison of percentage of subjects who test positive for COVID-19 spike protein antibodies based on disease modifying treatment;
Correlation of COVID-19 spike protein antibodies with B and T cell levels and immunoglobulins | 4-6 weeks
  Correlation of COVID-19 spike antibody presence and levels based on B and T cell subsets and overall immune globulin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Guarnaccia, MD, Principal Investigator — Griffin Hospital; Frederick Browne, MD, Principal Investigator — Griffin Hospital
Locations (1):
- Griffin Hospital, Derby, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified requests for IPD that underlie results in a publication will be made available to other researchers upon requests sent to the study PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be shared upon request following publication of our findings.
Access Criteria: The study PI will review and address requests for IPD.

REFERENCES:
- [Background] Parakkal D, Wooseob K, Paley MA, et al. Glucocorticoids and B Cell Depleting Agents Substantially Impair Immunogenicity of mRNA Vaccines to SARS-CoV-2 medRxiv 2021.04.05.21254656
- [Background] Boyarsky BJ, Werbel WA, Avery RK, Tobian AAR, Massie AB, Segev DL, Garonzik-Wang JM. Antibody Response to 2-Dose SARS-CoV-2 mRNA Vaccine Series in Solid Organ Transplant Recipients. JAMA. 2021 Jun 1;325(21):2204-2206. doi: 10.1001/jama.2021.7489. PMID 33950155
- [Background] Kennedy NA, Lin S, Goodhand JR, Chanchlani N, Hamilton B, Bewshea C, Nice R, Chee D, Cummings JF, Fraser A, Irving PM, Kamperidis N, Kok KB, Lamb CA, Macdonald J, Mehta S, Pollok RC, Raine T, Smith PJ, Verma AM, Jochum S, McDonald TJ, Sebastian S, Lees CW, Powell N, Ahmad T; Contributors to the CLARITY IBD study. Infliximab is associated with attenuated immunogenicity to BNT162b2 and ChAdOx1 nCoV-19 SARS-CoV-2 vaccines in patients with IBD. Gut. 2021 Oct;70(10):1884-1893. doi: 10.1136/gutjnl-2021-324789. Epub 2021 Apr 26. PMID 33903149
- [Background] Wu GF, Alvarez E. The immunopathophysiology of multiple sclerosis. Neurol Clin. 2011 May;29(2):257-78. doi: 10.1016/j.ncl.2010.12.009. PMID 21439440
- [Background] Popescu BF, Pirko I, Lucchinetti CF. Pathology of multiple sclerosis: where do we stand? Continuum (Minneap Minn). 2013 Aug;19(4 Multiple Sclerosis):901-21. doi: 10.1212/01.CON.0000433291.23091.65. PMID 23917093
- [Background] Weissert R. The immune pathogenesis of multiple sclerosis. J Neuroimmune Pharmacol. 2013 Sep;8(4):857-66. doi: 10.1007/s11481-013-9467-3. Epub 2013 May 10. PMID 23660832
- [Background] Doshi A, Chataway J. Multiple sclerosis, a treatable disease. Clin Med (Lond). 2016 Dec;16(Suppl 6):s53-s59. doi: 10.7861/clinmedicine.16-6-s53. PMID 27956442
- [Background] Zheng C, Kar I, Chen CK, Sau C, Woodson S, Serra A, Abboud H. Multiple Sclerosis Disease-Modifying Therapy and the COVID-19 Pandemic: Implications on the Risk of Infection and Future Vaccination. CNS Drugs. 2020 Sep;34(9):879-896. doi: 10.1007/s40263-020-00756-y. PMID 32780300
- [Background] Ciotti JR, Valtcheva MV, Cross AH. Effects of MS disease-modifying therapies on responses to vaccinations: A review. Mult Scler Relat Disord. 2020 Oct;45:102439. doi: 10.1016/j.msard.2020.102439. Epub 2020 Aug 1. PMID 32769063
- [Background] Brownlee WJ, Altmann DR, Prados F, Miszkiel KA, Eshaghi A, Gandini Wheeler-Kingshott CAM, Barkhof F, Ciccarelli O. Early imaging predictors of long-term outcomes in relapse-onset multiple sclerosis. Brain. 2019 Aug 1;142(8):2276-2287. doi: 10.1093/brain/awz156. PMID 31342055
- [Background] Altmann DM, Douek DC, Boyton RJ. What policy makers need to know about COVID-19 protective immunity. Lancet. 2020 May 16;395(10236):1527-1529. doi: 10.1016/S0140-6736(20)30985-5. Epub 2020 Apr 27. No abstract available. PMID 32353328
- [Background] Lurie N, Saville M, Hatchett R, Halton J. Developing Covid-19 Vaccines at Pandemic Speed. N Engl J Med. 2020 May 21;382(21):1969-1973. doi: 10.1056/NEJMp2005630. Epub 2020 Mar 30. No abstract available. PMID 32227757
- [Background] Karpinski TM, Ozarowski M, Seremak-Mrozikiewicz A, Wolski H, Wlodkowic D. The 2020 race towards SARS-CoV-2 specific vaccines. Theranostics. 2021 Jan 1;11(4):1690-1702. doi: 10.7150/thno.53691. eCollection 2021. PMID 33408775
- [Background] Kandimalla R, John A, Abburi C, Vallamkondu J, Reddy PH. Current Status of Multiple Drug Molecules, and Vaccines: An Update in SARS-CoV-2 Therapeutics. Mol Neurobiol. 2020 Oct;57(10):4106-4116. doi: 10.1007/s12035-020-02022-0. Epub 2020 Jul 15. PMID 32671688
- [Background] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] Sadoff J, Gray G, Vandebosch A, Cardenas V, Shukarev G, Grinsztejn B, Goepfert PA, Truyers C, Fennema H, Spiessens B, Offergeld K, Scheper G, Taylor KL, Robb ML, Treanor J, Barouch DH, Stoddard J, Ryser MF, Marovich MA, Neuzil KM, Corey L, Cauwenberghs N, Tanner T, Hardt K, Ruiz-Guinazu J, Le Gars M, Schuitemaker H, Van Hoof J, Struyf F, Douoguih M; ENSEMBLE Study Group. Safety and Efficacy of Single-Dose Ad26.COV2.S Vaccine against Covid-19. N Engl J Med. 2021 Jun 10;384(23):2187-2201. doi: 10.1056/NEJMoa2101544. Epub 2021 Apr 21. PMID 33882225
- [Background] Mohn N, Konen FF, Pul R, Kleinschnitz C, Pruss H, Witte T, Stangel M, Skripuletz T. Experience in Multiple Sclerosis Patients with COVID-19 and Disease-Modifying Therapies: A Review of 873 Published Cases. J Clin Med. 2020 Dec 16;9(12):4067. doi: 10.3390/jcm9124067. PMID 33339436
- [Background] Pinar Morales R, Ramirez Rivas MA, Barrero Hernandez FJ. SARS-CoV-2 infection and seroprevalence in patients with multiple sclerosis. Neurologia (Engl Ed). 2021 Nov-Dec;36(9):698-703. doi: 10.1016/j.nrleng.2021.03.002. Epub 2021 Jun 1. PMID 34103271
- [Background] Giovannoni G. Anti-CD20 immunosuppressive disease-modifying therapies and COVID-19. Mult Scler Relat Disord. 2020 Jun;41:102135. doi: 10.1016/j.msard.2020.102135. Epub 2020 Apr 18. No abstract available. PMID 32339915
- [Background] Sharifian-Dorche M, Sahraian MA, Fadda G, Osherov M, Sharifian-Dorche A, Karaminia M, Saveriano AW, La Piana R, Antel JP, Giacomini PS. COVID-19 and disease-modifying therapies in patients with demyelinating diseases of the central nervous system: A systematic review. Mult Scler Relat Disord. 2021 May;50:102800. doi: 10.1016/j.msard.2021.102800. Epub 2021 Jan 29. PMID 33578206
- [Background] Langer-Gould A, Smith JB, Li BH; KPSC MS Specialist Group. Multiple sclerosis, rituximab, and COVID-19. Ann Clin Transl Neurol. 2021 Apr;8(4):938-943. doi: 10.1002/acn3.51342. Epub 2021 Mar 30. PMID 33783140
- [Background] Kister I, Krogsgaard M, Mulligan MJ, Patskovsky Y, Voloshyna I, Ferstler N, Zhovtis Ryerson L, Curtin R, Kim J, Tardio E, Rimler Z, Sherman K, Samanovic-Golden M, Cornelius A, Lieberman D, Solis S, Pedotti R, Raposo C, Priest J, Hawker K, Silverman GJ. Preliminary Results of Ongoing, Prospective Study of Antibody and TCell Responses to SARS-CoV-2 in Patients With MS on Ocrelizumab or Other Disease-Modifying Therapies. Presented at the 73rd Congress of the American Academy of Neurology (AAN) Virtual 2021; 17-22 April 2021. P15.014
- [Background] Bar-Or A, Calkwood JC, Chognot C, Evershed J, Fox EJ, Herman A, Manfrini M, McNamara J, Robertson DS, Stokmaier D, Wendt JK, Winthrop KL, Traboulsee A. Effect of ocrelizumab on vaccine responses in patients with multiple sclerosis: The VELOCE study. Neurology. 2020 Oct 6;95(14):e1999-e2008. doi: 10.1212/WNL.0000000000010380. Epub 2020 Jul 29. PMID 32727835
- [Background] Epstein DJ, Dunn J, Deresinski S. Infectious Complications of Multiple Sclerosis Therapies: Implications for Screening, Prophylaxis, and Management. Open Forum Infect Dis. 2018 Jul 16;5(8):ofy174. doi: 10.1093/ofid/ofy174. eCollection 2018 Aug. PMID 30094293
- [Background] Winkelmann A, Loebermann M, Reisinger EC, Hartung HP, Zettl UK. Disease-modifying therapies and infectious risks in multiple sclerosis. Nat Rev Neurol. 2016 Apr;12(4):217-33. doi: 10.1038/nrneurol.2016.21. Epub 2016 Mar 4. PMID 26943779
- [Background] Achiron A, Mandel M, Dreyer-Alster S, Harari G, Magalashvili D, Sonis P, Dolev M, Menascu S, Flechter S, Falb R, Gurevich M. Author response to: Correspondence to humoral immune response to COVID-19 mRNA vaccine in patients with multiple sclerosis treated with high-efficacy disease-modifying therapies. Ther Adv Neurol Disord. 2021 May 29;14:17562864211020082. doi: 10.1177/17562864211020082. eCollection 2021. No abstract available. PMID 34104221
- [Background] Doria-Rose N, Suthar MS, Makowski M, O'Connell S, McDermott AB, Flach B, Ledgerwood JE, Mascola JR, Graham BS, Lin BC, O'Dell S, Schmidt SD, Widge AT, Edara VV, Anderson EJ, Lai L, Floyd K, Rouphael NG, Zarnitsyna V, Roberts PC, Makhene M, Buchanan W, Luke CJ, Beigel JH, Jackson LA, Neuzil KM, Bennett H, Leav B, Albert J, Kunwar P; mRNA-1273 Study Group. Antibody Persistence through 6 Months after the Second Dose of mRNA-1273 Vaccine for Covid-19. N Engl J Med. 2021 Jun 10;384(23):2259-2261. doi: 10.1056/NEJMc2103916. Epub 2021 Apr 6. No abstract available. PMID 33822494
- [Background] Spencer AJ, McKay PF, Belij-Rammerstorfer S, Ulaszewska M, Bissett CD, Hu K, Samnuan K, Blakney AK, Wright D, Sharpe HR, Gilbride C, Truby A, Allen ER, Gilbert SC, Shattock RJ, Lambe T. Heterologous vaccination regimens with self-amplifying RNA and adenoviral COVID vaccines induce robust immune responses in mice. Nat Commun. 2021 May 17;12(1):2893. doi: 10.1038/s41467-021-23173-1. PMID 34001897
- [Background] The combined use of AstraZeneca and Pfizer vaccines against SARS-CoV-2 offers a powerful immune response (isciii.es). https://www.isciii.es/Noticias/Noticias/Paginas/Noticias/Presentaci%c3%b3n-resultados-preliminares-CombivacS.aspx
- [Background] Shaw RH, Stuart A, Greenland M, Liu X, Nguyen Van-Tam JS, Snape MD; Com-COV Study Group. Heterologous prime-boost COVID-19 vaccination: initial reactogenicity data. Lancet. 2021 May 29;397(10289):2043-2046. doi: 10.1016/S0140-6736(21)01115-6. Epub 2021 May 12. No abstract available. PMID 33991480
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977